CLINICAL TRIAL: NCT06963905
Title: Phase Ib Randomized Open-label Trial of Sacituzumab Govitecan Plus Nivolumab or Sacituzumab Govitecan Plus Nivolumab and Relatlimab as Second-line Therapy for PD-L1 Positive Metastatic Triple Negative Breast Cancer
Brief Title: Saci Nivo Rela for TNBC
Acronym: SIMONE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Adriana Kahn, Assistant Professor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037105
Record Dates: First submitted 2025-04-02; First posted 2025-05-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Triple-negative Breast Cancer
Keywords: sacituzumab govitecan; PD-L1
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Nivolumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Sacituzumab govitecan plus a fixed dose combination of nivolumab and relatlimab
  Interventions: Drug: Relatlimab FDC + Nivolumab; Drug: Sacituzumab Govitecan (SG)
- Arm B (Active Comparator): Sacituzumab Govitecan plus nivolumab
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Nivolumab

INTERVENTIONS:
Drug: Relatlimab FDC + Nivolumab — Relatlimab: 360 IV Q3W (Dose level 1) and 120mg IV Q3W (Dose level -1) Nivolumab: 360mg IV Q3W
  Arms: Arm A
Drug: Sacituzumab Govitecan (SG) — 10 mg/kg IV D1 & D8 every 21-day cycles (Dose level 1); 7.5 mg/kg IV D1 & D8 every 21-day cycles (Dose level -1); 5 mg/kg IV D1 & D8 every 21-day cycles 21-day cycles (Dose level -2)
Drug: Nivolumab — 360mg IV Q3W
  Arms: Arm B

SUMMARY:
This is a randomized, open-label, phase Ib study to assess safety and efficacy of sacituzumab govitecan plus nivolumab or sacituzumab govitecan plus a fixed dose combination of nivolumab and relatlimab in patients with programmed cell death-ligand 1 (PD-L1) positive (defined by combined positive score >10), metastatic, triple negative breast cancer on routine testing with one prior line of cytotoxic chemotherapy with pembrolizumab in the metastatic setting. The study treatment will be continued until the progression of disease, unacceptable toxicity, death, or withdrawal of consent for any reason.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase Ib study to assess safety and efficacy of sacituzumab govitecan plus nivolumab or sacituzumab govitecan plus a fixed dose combination of nivolumab and relatlimab in patients with programmed cell death-ligand 1 (PD-L1) positive (defined by combined positive score >10), metastatic, triple negative breast cancer on routine testing with one prior line of cytotoxic chemotherapy with pembrolizumab in the metastatic setting. The study treatment will be continued until the progression of disease, unacceptable toxicity, death, or withdrawal of consent for any reason. Patients will be followed up for up to two years. Their safety will be monitored, and tumor response will be regularly evaluated by RECIST 1.1 criteria every nine weeks. The primary endpoint includes safety as the incidence of dose-limiting toxicities (DLT) in three weeks after C1D1. Secondary endpoints include overall response rate (defined as either complete response or partial response), duration of response, clinical benefit rate, progression free survival, and safety (TEAE) with sacituzumab govitecan plus nivolumab or sacituzumab govitecan plus nivolumab + relatlimab FDC. Exploratory endpoints include overall survival, and biomarkers of prediction of response will be also evaluated. There will be a 135-day (+7 days) follow-up visit after the last study treatment administration or before starting a new anticancer treatment, whichever occurs first, followed by long-term/survival chart review follow-up every three months (±14 days) from the date of the 135-day (+7 days) follow-up visit for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date an IRB approved ICF before the performance of any study specific procedures or tests.
2. Participants 18 years or older.
3. Pathologically documented breast cancer that:

   1. Is defined as unresectable/metastatic disease.
   2. Is Human Epidermal Growth Factor Receptor 2 (HER2)-negative, defined as HER2- immunohistochemistry (IHC) 0, 1+ or 2+ ISH negative, and estrogen receptor (ER)- and progesterone receptor (PgR)- negative, both defined as IHC <10%
   3. PD-L1 positive disease as per IHC via CPS > 10 by IHC (defined by the number of PD-L1 staining cells [tumor cells, lymphocytes, macrophages] divided by the total number of viable tumor cells, multiplied by 100) via FDA-approved SP263 assay..
   4. Has been treated with up to one line of systemic cytotoxic chemotherapy with pembrolizumab in the metastatic setting. If recurrence occurred within six months of (neo)adjuvant chemotherapy, (neo)adjuvant chemotherapy would count as one line of therapy.
   5. Prior immune checkpoint inhibition with systemic chemotherapy is required in either neo(adjuvant) or metastatic settings
   6. Prior targeted therapies (e.g., olaparib, or others upon discussion with study sponsor-investigator) do not count as systemic cytotoxic chemotherapy lines and are unlimited prior to enrolment.
4. Documented radiologic progression (during or after most recent treatment) or intolerance to prior line of therapy regardless of prior response with subsequent medical need for change of therapy.
5. Must have an adequate archival tumor sample <3 years old available for assessment of PD-L1 status by IHC via CPS. If archival tissue is not available or inadequate for assessment (e.g., decalcified bone, cytology, or other), a fresh biopsy is required on enrolment.
6. Presence or absence of measurable lesion based on computed tomography (CT) or MRI per modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1 are both allowed.
7. ECOG PS 0 or 1.
8. Left ventricular ejection fraction (LVEF) ≥50% within 6 months prior to enrolment.
9. Adequate laboratory parameters (table 1) within 14 days from C1D1
10. Adequate contraception when indicated (table 2), such as:

    1. Evidence of post-menopausal status or negative serum pregnancy test for participants of childbearing potential who are sexually active with a non-sterilized male partner.
    2. For participants of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of study drugs.
    3. Participants of childbearing potential are defined as those who are not surgically sterile (i.e., underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Participants will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
    4. Participants of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in table 3, from the time of screening and must agree to continue using such precautions for seven months after the last dose of study drugs.
    5. Female participants must refrain from breastfeeding while on study and for seven months after the last dose of study drugs.
    6. Female participants must not donate, or retrieve for their own use, ova from the time of enrolment and throughout the study treatment period, and for at least seven months after the final study drug administration. Preservation of ova may be considered prior to enrolment in this study.
    7. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the participant's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
    8. Non-sterilized male participants who are sexually active with a female partner of childbearing potential must use a condom from screening to five months after the final dose of study drugs.
    9. Male participants should refrain from fathering a child or freezing or donating sperm from the time of enrolment, throughout the study, and for five months after the last dose of study drugs. Preservation of sperm should be considered prior to enrolment in this study.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Participants who are pregnant or lactating.
2. Participants of childbearing potential or fertile men unwilling to use effective contraception.
3. Certain prior comorbidities, such as:

   1. Concomitant metastatic disease from other primary tumors.
   2. Known history of unstable angina, MI, or CHF present within six months of randomization or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy.
   3. History of myocarditis.
   4. Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within six months of randomization.
   5. History of (non-infectious) pneumonitis or interstitial pulmonary disease that required steroids for more than 28 consecutive days or has current pneumonitis or interstitial pulmonary disease.
   6. Prior history of GI perforation within six months of randomization.
   7. Has an uncontrolled infection requiring current IV antibiotics, antivirals, or antifungals.
   8. Has known human immunodeficiency virus (HIV) infection with detectable viral load or CD4 count < 200 cells per cubic millimeter or active hepatitis B (HBsAg positive) or C (HCV positive RNA) infection.
   9. Any active autoimmune, connective tissue or inflammatory disorders that required active immunomodulatory or corticosteroid treatments in the two years prior to study enrolment. Participants with active autoimmune diseases may enroll with the following conditions: type 1 diabetes mellitus; hypothyroidism only requiring hormone replacement; skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
4. Certain central nervous system conditions, such as:

   1. Has currently untreated spinal cord compression.
   2. Has clinically active central nervous system metastases, defined as symptomatic, or requiring therapy with corticosteroids to control associated symptoms.
   3. Participants with clinically asymptomatic brain metastases not requiring corticosteroids and seizure-free for more than 30 days with or without prior local therapy administration (surgery and/or radiation therapy) may be included in the study.
   4. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
5. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade ≤1 or baseline. Participants with chronic grade 2 toxicities may be eligible per the discretion of the investigator (e.g., grade 2 chemotherapy-induced neuropathy, fatigue, residual endocrinopathies from use of immunotherapy such as hypothyroidism/hyperthyroidism, type 1 diabetes, hyperglycemia, adrenal insufficiency, adrenalitis, skin hypopigmentation (vitiligo)).
6. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
7. Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
8. Participants must not have had prior treatment with relatlimab or any other LAG-3 targeted agent, as well as no prior SG.
9. Substance abuse, medical conditions, social, familial, or geographical factors that would, in the opinion of the investigator, increase the safety risk to the participant or interfere with the participant's participation in the clinical study or evaluation of the clinical study results despite best use of locally and community available resources.
10. Adequate washout period from prior therapies before C1D1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities in patients treated with sacituzumab govitecan combinations | Three weeks post-Cycle 1 Day 1 (each cycle is 21 days)
  The primary outcome measure is the incidence of dose-limiting toxicities (DLTs) observed three weeks after the first cycle of treatment with sacituzumab govitecan in combination with nivolumab, or sacituzumab govitecan in combination with nivolumab and relatlimab fixed-dose combination in patients with advanced triple-negative breast cancer in the second-line setting. The assessment will include the frequency and severity of DLTs to evaluate the safety and tolerability of the treatment regimens.

SECONDARY OUTCOMES:
Time to response in patients treated with sacituzumab govitecan combinations | At baseline (Week 0), followed by assessments every 9 weeks (Weeks 9, 18, 27, 36, etc.). The final assessment will take place at the end of the trial, during the last follow-up visit, which will occur 4 weeks post-treatment or upon study completion
  Time to Response is defined as the time from the initiation of treatment to the first documentation of a complete response or partial response in patients with advanced TNBC in the second-line setting. This outcome measure will assess the efficacy of sacituzumab govitecan in combination with nivolumab, or sacituzumab govitecan in combination with nivolumab and relatlimab FDC, by measuring how quickly patients respond to the therapy..
Overall response rate in patients treated with sacituzumab govitecan combinations | At baseline (Week 0), followed by assessments every 9 weeks (Weeks 9, 18, 27, 36, etc.). The final assessment will take place at the end of the trial, during the last follow-up visit, which will occur 4 weeks post-treatment or upon study completion
  The Overall Response Rate is defined as the proportion of patients with advanced triple-negative breast cancer in the second-line setting who achieve either a complete response or partial response according to the RECIST version 1.1. The ORR will be assessed in patients receiving sacituzumab govitecan combined with nivolumab, or sacituzumab govitecan combined with nivolumab and relatlimab fixed-dose combination (FDC). This outcome measure aims to evaluate the preliminary efficacy of the treatment regimens.
Duration of response in patients treated with sacituzumab govitecan combinations | At baseline (Week 0), followed by assessments every 9 weeks (Weeks 9, 18, 27, 36, etc.). The final assessment will take place at the end of the trial, during the last follow-up visit, which will occur 4 weeks post-treatment or upon study completion
  The Duration of Response is defined as the time from the first documentation of a complete response or partial response until the time of disease progression or death from any cause, whichever occurs first. This measure will be evaluated in patients with advanced TNBC in the second-line setting who respond to treatment with sacituzumab govitecan plus nivolumab, or sacituzumab govitecan plus nivolumab and relatlimab FDC. The objective is to determine the sustainability of the responses induced by the treatment combinations.
Clinical benefit rate in patients treated with sacituzumab govitecan combinations | At baseline (Week 0), followed by assessments every 9 weeks (Weeks 9, 18, 27, 36, etc.). The final assessment will take place at the end of the trial, during the last follow-up visit, which will occur 4 weeks post-treatment or upon study completion
  The Clinical Benefit Rate is defined as the proportion of patients who achieve a complete response, partial response, or stable disease for at least 6 months, according to RECIST version 1.1. This measure will be assessed in patients with advanced TNBC in the second-line setting undergoing treatment with sacituzumab govitecan plus nivolumab, or sacituzumab govitecan plus nivolumab and relatlimab FDC. The CBR will help determine the overall efficacy and potential benefit of the treatment regimens.
Progression free survival in patients treated with sacituzumab govitecan combinations | At baseline (Week 0), followed by assessments every 9 weeks (Weeks 9, 18, 27, 36, etc.). The final assessment will take place at the end of the trial, during the last follow-up visit, which will occur 4 weeks post-treatment or upon study completion
  Progression-Free Survival is defined as the time from the start of treatment to the occurrence of disease progression or death from any cause, whichever occurs first. Disease progression will be assessed according to the RECIST version 1.1. This outcome measure will evaluate the preliminary efficacy of the treatment regimens involving sacituzumab govitecan in combination with nivolumab, or sacituzumab govitecan in combination with nivolumab and relatlimab fixed-dose combination (FDC) in patients with advanced triple-negative breast cancer (TNBC) in the second-line setting. The intent is to determine how effectively these treatment combinations can delay disease progression and extend the time patients remain progression-free.
Incidence of adverse events in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The incidence of adverse events will be assessed in patients with advanced triple-negative breast cancer in the second-line setting receiving treatment with sacituzumab govitecan plus nivolumab, or sacituzumab govitecan plus nivolumab and relatlimab fixed-dose combination (FDC). Adverse events will be recorded and graded according to NCI CTCAE version 5.0.
Frequency of serious adverse events in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The frequency of serious adverse events will be monitored and documented in patients treated with sacituzumab govitecan in combination with nivolumab, or sacituzumab govitecan in combination with nivolumab and relatlimab FDC. SAEs will be classified and graded according to the NCI CTCAE version 5.0 criteria.
Incidence of Treatment-Emergent Adverse Events in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  Treatment-emergent adverse events will be defined and assessed as any adverse events that arise following the initiation of treatment with sacituzumab govitecan plus nivolumab, or sacituzumab govitecan plus nivolumab and relatlimab FDC. TEAEs will be graded according to the NCI CTCAE version 5.0 criteria.
Incidence of Adverse Events of Special Interest in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The incidence of adverse events of special interest will be recorded and evaluated in patients receiving treatment with sacituzumab govitecan combinations. AESIs will include specific adverse events deemed critical based on the known safety profile of the drugs, and will be graded according to the NCI CTCAE version 5.0 criteria.
Incidence of Immune-Mediated Adverse Events in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The occurrence of immune-mediated adverse events will be monitored in patients treated with sacituzumab govitecan in combination with nivolumab, or sacituzumab govitecan in combination with nivolumab and relatlimab FDC. imAEs will be assessed and graded according to NCI CTCAE version 5.0 criteria to describe the immune-related safety profile of the treatment regimens.
Rate of Treatment Discontinuation Due to Adverse Events in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The rate at which patients discontinue treatment due to adverse events will be assessed. This measure will monitor the proportion of patients with advanced TNBC in the second-line setting who cease treatment with sacituzumab govitecan combinations due to AEs. AEs leading to discontinuation will be documented and graded according to NCI CTCAE version 5.0 criteria.
Changes in ECOG Performance Status in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle and at the last follow up visit, 30 days after the last treatment cycle or upon study completion
  The changes in Eastern Cooperative Oncology Group (ECOG) Performance Status will be evaluated at baseline and periodically during treatment to assess the impact of sacituzumab govitecan combinations on patients' functional status. The ECOG Performance Status scale will be utilized to categorize patient performance levels.
Electrocardiogram abnormalities in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle
  Electrocardiogram (ECG) assessments will be conducted to monitor for any treatment-related cardiac abnormalities in patients receiving sacituzumab govitecan combinations. Any significant ECG changes and their clinical relevance will be documented.
Echocardiogram findings in patients treated with sacituzumab govitecan combinations | Days 1 and 8 of every 21-day cycle
  Echocardiogram (ECHO) assessments will be performed to evaluate cardiac function and detect any cardiotoxicity associated with sacituzumab govitecan plus nivolumab, or sacituzumab govitecan plus nivolumab and relatlimab FDC. ECHO findings will be analyzed for any significant changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Kahn, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No